CLINICAL TRIAL: NCT05567809
Title: DEFINE-TAVR (Defining Exercise Hemodynamics and Function After Transcatheter Aortic Valve Replacement) Study
Brief Title: Defining Exercise Hemodynamics and Function After Transcatheter Aortic Valve Replacement (DEFINE-TAVR) Study.
Acronym: DEFINE-TAVR
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Anteris Technologies Corporation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2000033211; YSI-002 (Other: Yale)
Record Dates: First submitted 2022-09-28; First posted 2022-10-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to help understand how the replacement valve functions over time, both at rest and during exercise.

DETAILED DESCRIPTION:
The objective of this single-center registry is to evaluate prosthetic valve hemodynamics and function over time in patients undergoing clinically indicated transcatheter aortic valve replacement (TAVR) for symptomatic severe aortic stenosis. Specific goals include:

* Describe valve hemodynamics at rest (baseline, post-procedure, 30 days, 1 year) and with exercise (at 30 days and 1 year) after TAVR implantation to define valve function and hemodynamics over time.
* Compare valve hemodynamics and function at rest and exercise between self-expanding and balloon expandable valves.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female ≥18 years of age
* Clinically indicated for TAVR
* Aortic annular size measures 21-25 mm diameter based on pre-procedure Computed Tomography Angiography (CTA)
* Able to exercise and, in the judgment of the investigator, is likely to be physically able to comply with the protocol requirements regarding exercise echocardiography
* Willing to comply with protocol-specified follow-up evaluations
* The participant or legally authorized representative, has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

* Previously implanted prosthetic aortic valve (i.e., planned valve-in-valve TAVR)
* Known mental or physical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation, or is associated with a life expectancy of less than one year
* Left ventricular ejection fraction (LVEF) <35%
* Presenting with cardiogenic shock at the time of the index procedure
* Planned to undergo any cardiac surgical procedure in the following 12 months
* The index procedure results in an unsuccessful TAVR, defined as procedural major adverse events (death, disabling stroke, or life-threatening or disabling bleeding), need for a second prosthesis implant, or conversion to emergent surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A minimum of 50 and up to 100 adults presenting with symptomatic severe aortic stenosis referred for clinically indicated TAVR at Yale New Haven Hospital who meet all eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
TransAortic Valve Gradient during exercise at 12 months post-TAVR | 12 months post-TAVR
  TransAortic Valve Gradient (mmHg) during exercise as assessed by the Echocardiographic Core Laboratory and summarized as peak and mean.

SECONDARY OUTCOMES:
Change in valve cusp thickness at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in valve cusp thickness (mm) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in valve mobility at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in valve mobility at rest assessed using echocardiogram reported as absolute values and as changes.
Change in paravalvular leak at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in paravalvular leak at rest assessed using echocardiogram reported as absolute values and as changes.
Change in coefficient of contraction Effective Orifice Area (EOA)/Geometric Orifice Area (GOA) at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in coefficient of contraction EOA/GOA at rest assessed using echocardiogram reported as absolute values and as changes.
Change in Dimensionless Velocity Index (DVI) at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in DVI at rest assessed using echocardiogram reported as absolute values and as changes.
Change in energy loss coefficient at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in energy loss coefficient at rest assessed using echocardiogram reported as absolute values and as changes.
Change in EOA at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in EOA (cm2) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in aortic valve gradient (peak and mean) at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in aortic valve gradient (mmHg) (peak and mean) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in aortic valve velocity (peak and mean) at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in aortic valve velocity (m/s) (peak and mean) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in Left Ventricle (LV) remodeling at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in LV remodeling at rest assessed using echocardiogram reported as absolute values and as changes.
Change in leaflet thickening at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in leaflet thickening at rest assessed using echocardiogram reported as absolute values and as changes.
Change in coaptation length at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in coaptation length (mm) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in LV thickness at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in LV thickness (cm) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in LV Global Longitudinal Strain at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in LV Global Longitudinal Strain (%) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in Right Ventricular (RV) systolic velocity at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in RV systolic velocity (cm/s) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in RV systolic pressure (RVSP) at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in RVSP (mmHg) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) at rest | baseline, during hospitalization approximatively 3 days, 30 days, and 12 months post-TAVR
  Change in TAPSE (mm) at rest assessed using echocardiogram reported as absolute values and as changes.
Change in aortic valve gradient (peak and mean) with exercise | 30 days, and 12 months post-TAVR
  Change in gradient (mmHg) (peak and mean) with exercise assessed using echocardiogram reported as absolute values and as changes.
Change in aortic valve velocity (peak and mean) with exercise | 30 days and 12 months post-TAVR
  Change in aortic valve velocity (m/s) (peak and mean) with exercise assessed using echocardiogram reported as absolute values and as changes.
Change in DVI with exercise | 30 days and 12 months post-TAVR
  Change in DVI with exercise assessed using echocardiogram reported as absolute values and as changes.
Change in EOA with exercise | 30 days and 12 months post-TAVR
  Change in EOA (cm2) with exercise assessed using echocardiogram reported as absolute values and as changes.
Change in RVSP with exercise | 30 days and 12 months post-TAVR
  Change in RVSP (mmHg) with exercise assessed using echocardiogram reported as absolute values and as changes.
Change in exercise duration | 30 days and 12 months post-TAVR
  Change in exercise duration (min) reported as absolute values and as changes.
Change in LV Global Longitudinal Strain with exercise | 30 days and 12 months post-TAVR
  Change in LV Global Longitudinal Strain (%) with exercise assessed using echocardiogram reported as absolute values and as changes.
TAVR Device Success (Valve Academic Research Consortium [VARC]-defined) | during hospitalization approximatively 3 days
  TAVR Device Success evaluated post-procedure/pre-discharge during hospitalization approximatively 3 days, defined as: absence of procedural mortality AND correct positioning of a single prosthetic heart valve into the proper anatomical location AND intended performance of the prosthetic heart valve (defined as no prosthesis-patient mismatch [VARC-defined] and mean aortic valve gradient <20 mm Hg or peak velocity <3 m/s, AND no moderate or severe prosthetic valve regurgitation [VARC-defined] [site and Core Laboratory-reported].
Composite Safety Endpoints (VARC-3 defined) | 30 days and 12 months post-TAVR
  Composite safety endpoint reported as a proportion of participants who died or experienced neurological events or life-threatening bleeding or acute kidney injury or coronary artery obstruction requiring intervention or major vascular complications or valve-related dysfunction requiring repeat procedure evaluated at 30 days and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Vora, MD, Principal Investigator — Yale University; Alexandra J Lansky, MD, Study Chair — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No